CLINICAL TRIAL: NCT06956664
Title: Comparative Efficacy of Physiotherapeutic Exercise Regimens Implemented After Caudal Epidural Steroid Injection
Brief Title: Exercise Therapy After Caudal Epidural Steroid Injection
Acronym: CAPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ceyhun Türkmen, Assoc. Prof. Dr., Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ec5190f6baf84e82
Record Dates: First submitted 2025-04-23; First posted 2025-05-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Intervertebral Disc Displacement; Low Back Pain; Radiculopathy
Keywords: Caudal Epidural Injection; Low Back Pain; Exercise Therapy; Aerobic Exercise; Core Stabilization
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain; Radiculopathy

STUDY DESIGN:
Intervention Model Description: Randomised, three-arm, parallel-group trial. Participants are allocated 1:1:1 to one of the following interventions delivered for six weeks:
  Conventional physiotherapy alone (heat, ultrasound, TENS)
  Conventional physiotherapy + aerobic treadmill exercise
  Conventional physiotherapy + progressive core-stabilisation exercise Groups receive their assigned programme concurrently for the full study duration; no crossover or adaptive sequencing is planned.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The treating physiotherapists and participants cannot be blinded because the nature of the exercise programmes is overt. However, (i) outcome assessors who perform all baseline and follow-up measurements and (ii) the trial statistician responsible for primary analyses will remain unaware of group allocation. Randomisation codes are stored in sealed, opaque envelopes by a study coordinator not involved in assessment or analysis, and participants are reminded not to disclose their exercise group during evaluations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy (Active Comparator): Other: Conventional Physiotherapy (moist heat, therapeutic ultrasound, TENS)
  Interventions: Other: Conventional Physiotherapy
- Aerobic Exercise + Conventional Physiotherapy (Experimental): * Behavioral: Aerobic Exercise (treadmill walking)
  * Other: Conventional Physiotherapy
  Interventions: Other: Conventional Physiotherapy; Behavioral: Aerobic Exercise Programme
- Core-Stabilization Exercise + Conventional Physiotherapy (Experimental): * Behavioral: Core-Stabilisation Exercise
  * Other: Conventional Physiotherapy
  Interventions: Other: Conventional Physiotherapy; Behavioral: Core-Stabilization Exercise Programme

INTERVENTIONS:
Other: Conventional Physiotherapy — Standard physical-agent package delivered three times weekly for 6 weeks: 20 min moist hot-pack (≈70 °C hydrocollator packs); 5 min continuous therapeutic ultrasound (1 MHz, 1 W cm-²); 20 min biphasic TENS (100 Hz, 100 µs). Initiated 2 weeks after the caudal epidural steroid injection (CESI).
Behavioral: Aerobic Exercise Programme — Supervised treadmill walking three times weekly for 6 weeks: 5 min warm-up at ~40 % HR<sub>max</sub>; 10-25 min load at 55-80 % HR<sub>max</sub> (5 % weekly progression); 5 min cool-down. Heart-rate telemetry and Borg CR-10 used to titrate intensity. Starts 2 weeks post-CESI.
  Arms: Aerobic Exercise + Conventional Physiotherapy
Behavioral: Core-Stabilization Exercise Programme — Phased lumbopelvic motor-control regimen three times weekly for 6 weeks: Phase I isolated transversus abdominis/multifidus activation with pressure biofeedback; Phase II functional co-contraction with limb movements in quadruped, sitting, standing; Phase III dynamic tasks on Swiss-ball/BOSU with resistance. Progression requires pain ≤ 3/10 VAS and flawless technique. Begins 2 weeks post-CESI.
  Arms: Core-Stabilization Exercise + Conventional Physiotherapy

SUMMARY:
**Brief Summary**

Lumbar radicular pain arising from intervertebral disc herniation is commonly managed with a caudal epidural steroid injection (CESI), a minimally invasive procedure that delivers anti-inflammatory medication to the sacral hiatus. Although CESI affords short-term analgesia, a sizable proportion of patients continue to experience pain-related disability and diminished quality of life, underscoring the need for optimised post-injection rehabilitation.

This single-centre, three-arm, parallel-group randomised controlled trial will evaluate the comparative efficacy of two evidence-informed exercise paradigms-moderate-intensity aerobic training and progressive lumbopelvic stabilisation-when each is superimposed upon a standard physiotherapy package of heat, therapeutic ultrasound and transcutaneous electrical nerve stimulation (TENS). Forty-two adults (18-70 years) with MRI-confirmed lumbar disc herniation who have undergone CESI at Çankırı State Hospital will be randomly allocated (1:1:1) to one of the following six-week interventions, initiated two weeks post-injection and delivered thrice weekly under physiotherapist supervision:

1. Conventional physiotherapy alone (heat + ultrasound + TENS).
2. Conventional physiotherapy plus aerobic exercise (treadmill walking at 55-80 % of age-predicted maximal heart rate with structured warm-up/cool-down).
3. Conventional physiotherapy plus core-stabilisation exercise (phased activation of deep trunk musculature progressing to dynamic tasks on unstable surfaces).

Primary end-points are pain intensity (10 cm Visual Analogue Scale) and back-specific disability (Oswestry Disability Index). Secondary end-points include generic health-related quality of life (SF-12) and lumbar proprioceptive body awareness (Fremantle Back Awareness Questionnaire). Outcomes will be captured at baseline, post-intervention (6 weeks) and at 3- and 6-month follow-up to ascertain both immediate and sustained effects.

Study Question Does adjunctive aerobic or core-stabilisation exercise confer superior reductions in pain and disability, and greater gains in quality of life and body awareness, compared with conventional physiotherapy alone in adults following CESI for lumbar disc herniation?

It is hypothesised that both exercise approaches will yield clinically and statistically superior outcomes relative to standard care, with stabilisation training providing the most durable functional benefits. Findings are expected to refine post-CESI rehabilitation algorithms and inform evidence-based clinical guidance for physiotherapists managing lumbar disc pathology.

DETAILED DESCRIPTION:
Scientific Rationale and Background Caudal epidural steroid injection (CESI) is widely employed to attenuate lumbosacral radicular pain by delivering glucocorticoids into the sacral hiatus, thereby diminishing local biochemical inflammation around the affected nerve roots. While CESI frequently yields rapid analgesia, pain recurrence and activity limitation are common within three to six months, indicating that pharmacological attenuation of inflammation alone is insufficient to restore neuromuscular control and functional capacity. Emerging evidence suggests that structured exercise commenced shortly after CESI can exploit the "analgesic window" to retrain motor patterns, enhance spinal stability, and improve cardiovascular fitness-yet the optimal exercise paradigm remains unclear. Aerobic conditioning may promote anti-inflammatory myokine release and general de-conditioning reversal, whereas lumbopelvic stabilisation targets segmental control deficits and proprioceptive impairment-both recognised contributors to chronicity in lumbar disc pathology.

Study Design and Setting This is a single-centre, prospective, three-arm, parallel-group, superiority randomised controlled trial conducted at the Department of Physiotherapy, Çankırı State Hospital, Türkiye. Allocation (1:1:1) is computer-generated with permuted blocks of variable size; assignments are sealed in sequentially numbered opaque envelopes by an independent statistician to ensure allocation concealment. Outcome assessors and data analysts are blinded to group assignment. Interventions are delivered in a dedicated physiotherapy gymnasium under the supervision of senior musculoskeletal physiotherapists trained in study procedures.

Intervention Logic

Each participant receives a two-week "wash-in" period following CESI to permit stabilisation of acute pharmacodynamic effects. Thereafter, three arms are implemented over six weeks (18 supervised sessions):

1. Conventional Physiotherapy (control) - superficial moist heat (20 min, 70 °C hydrocollator packs), continuous ultrasound (1 MHz, 1.0 W cm-², 5 min), and biphasic TENS (100 Hz, 100 µs, 20 min).
2. Conventional Physiotherapy + Aerobic Exercise - identical modality package followed by treadmill walking at 55-80 % age-predicted HR_max with 5 min warm-up, 10-25 min load (weekly 5 % progression), and 5 min cool-down. Heart rate is telemetrically monitored; intensity is titrated using the Borg CR-10 scale and Tanaka equation (208-0.7·age).
3. Conventional Physiotherapy + Core-Stabilisation Exercise - modality package followed by a phased stabilisation protocol:

   * Phase I: isolated transversus abdominis and multifidus activation in supine/prone using pressure biofeedback (2 weeks).
   * Phase II: functional co-contraction with limb movements in quadruped, sitting, and standing (2 weeks).
   * Phase III: dynamic tasks on unstable surfaces (Swiss-ball, BOSU) incorporating resistance bands (2 weeks).

Progression criteria include pain ≤3/10 on VAS and flawless technique for ≥10 repetitions; repetitions, load, or surface instability are advanced by ~10 % weekly.

All participants receive a standardised education booklet on spine-sparing strategies and are advised to maintain normal activities.

Sample Size Justification Using an anticipated between-group effect size of d = 1.0 for pain reduction-derived from prior work on CESI-augmented exercise (Cohen's f = 0.5)-42 participants (14 per arm) provide 80 % power (α = 0.05, two-sided) to detect clinically important differences, allowing for 25 % attrition.

Data Management and Statistical Plan Data are entered into REDCap with double-entry verification. The primary analysis follows the intention-to-treat principle, employing linear mixed-effects models with random intercepts for participants, fixed effects for group, time, and their interaction, and baseline score as covariate. Missing data will be handled using restricted maximum likelihood under a missing-at-random assumption; sensitivity analyses will include multiple imputation. Secondary outcomes will be analysed similarly with Bonferroni-adjusted confidence intervals. Effect sizes (Hedges g) and minimal clinically important differences will be reported.

Safety Monitoring Adverse events-including exacerbation of radicular pain, hemodynamic instability during aerobic sessions, or procedure-related complications-are recorded at each visit. An independent physician adjudicates seriousness and relatedness; criteria for withdrawal include VAS ≥ 7 persisting >48 h or cardiovascular red-flags according to American College of Sports Medicine guidelines. A Data Safety Monitoring Sub-committee reviews unblinded safety reports quarterly.

*Knowledge Translation* Results will inform evidence-based guidelines on post-CESI rehabilitation, disseminated via peer-reviewed publication, conference presentation, and integration into continuing professional development modules for physiotherapists. De-identified datasets and analytic code will be deposited in an open repository within 12 months of primary outcome publication, aligning with FAIR data principles and UK Research Councils' open-science policy.

In summary, this rigorously designed trial seeks to delineate whether adjunctive aerobic or motor-control-oriented exercise offers superior and durable benefits over conventional modalities alone in the critical post-injection period for patients with lumbar disc herniation, thereby refining best-practice rehabilitation pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years.
* MRI-confirmed lumbar intervertebral disc herniation.
* Has received a caudal epidural steroid injection (CESI) within the past 2 weeks at Çankırı State Hospital.
* Low-back or leg pain intensity ≥ 3 cm on a 10-cm Visual Analogue Scale after the injection.
* Medically cleared for moderate aerobic and core-stabilisation exercise (no cardiac or orthopaedic contraindications).
* Able to attend supervised physiotherapy three times per week for six weeks.
* Willing and able to give written informed consent and to comply with study procedures.
* Sufficient Turkish literacy (minimum primary-school education) to complete questionnaires.

Exclusion Criteria:

* Uncontrolled systemic disease (e.g., poorly controlled diabetes mellitus, congestive heart failure, active hepatitis C or other significant liver disease).
* Neurological red flags such as myelopathy or cauda equina syndrome.
* Previous lumbar spine surgery at the affected disc level.
* Current pregnancy or planning pregnancy during the study period.
* Severe musculoskeletal, cardiovascular, or respiratory condition that precludes safe exercise participation.
* Use of systemic corticosteroids or opioid analgesics that cannot be stabilised for the duration of the trial.
* Ongoing litigation or workers' compensation claim related to low-back pain.
* Inability to communicate effectively with study staff or to follow instructions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (Numeric Rating Scale, 0-10) | Baseline; 6 weeks; 3 months; 6 months
  Unit of Measure: points on a 0-to-10 scale Description: 11-point Numeric Rating Scale; 0 = no pain, 10 = worst imaginable pain. Change from baseline will be calculated at each follow-up. Higher scores indicate worse pain.

SECONDARY OUTCOMES:
Change in Disability (Oswestry Disability Index, 0-100) | Baseline, 6 weeks, 3 months, 6 months
  Unit of Measure: percentage points (0-100) Description: Oswestry Disability Index v2.1a; higher scores denote greater disability. Change from baseline will be reported.
Change in Health-Related Quality of Life (SF-12 Physical Component, 0-100) | Baseline, 6 weeks, 3 months, 6 months
  Unit of Measure: points (0-100) Description: Short-Form-12 v2 Physical Component Summary (PCS); higher scores represent better quality of life.
Change in Health-Related Quality of Life (SF-12 Mental Component, 0-100) | Baseline; 6 weeks; 3 months; 6 months
  Short-Form-12 v2. Mental Component Summary (MCS) scores; higher values = better QoL. Change from baseline calculated for each follow-up.
Change in Lumbar Body Awareness (Fremantle Back Awareness Questionnaire, 0-36) | Baseline; 6 weeks; 3 months; 6 months
  Unit of Measure: points (0-36) Description: 9-item FreBAQ; higher scores reflect poorer body perception. Change from baseline reported.
Return-to-Work Days | Up to 6 months
  Unit of Measure: days Description: Self-reported calendar days from CESI to full resumption of habitual occupational duties. Lower values indicate faster return.

OTHER OUTCOMES:
Adverse Events Related to Exercise or CESI | Throughout 6-week intervention and 6-month follow-up
  Unit of Measure: number of participants with ≥1 event Description: Musculoskeletal, cardiovascular, or injection-related adverse events, coded per CTCAE v5.0. Both incidence and narrative description will be provided.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Çankırı Karatekin University, Çankırı
  - Çankırı State Hospital, Çankırı

IPD SHARING:
Plan to Share IPD: Yes
A de-identified participant-level dataset and accompanying data dictionary will be deposited in an open-access repository (e.g., Open Science Framework) within 12 months of publication of the primary results, accessible to qualified researchers under a CC-BY license.

REFERENCES:
- [Background] Zhang J, Zhang R, Wang Y, Dang X. Efficacy of epidural steroid injection in the treatment of sciatica secondary to lumbar disc herniation: a systematic review and meta-analysis. Front Neurol. 2024 May 22;15:1406504. doi: 10.3389/fneur.2024.1406504. eCollection 2024. PMID 38841695
- [Background] Yang H, Liu H, Li Z, Zhang K, Wang J, Wang H, Zheng Z. Low back pain associated with lumbar disc herniation: role of moderately degenerative disc and annulus fibrous tears. Int J Clin Exp Med. 2015 Feb 15;8(2):1634-44. eCollection 2015. PMID 25932092
- [Background] Yaman O, Guchkha A, Vaishya S, Zileli M, Zygourakis C, Oertel J. The role of conservative treatment in lumbar disc herniations: WFNS spine committee recommendations. World Neurosurg X. 2024 Feb 13;22:100277. doi: 10.1016/j.wnsx.2024.100277. eCollection 2024 Apr. PMID 38389961
- [Background] Yakut E, Duger T, Oksuz C, Yorukan S, Ureten K, Turan D, Frat T, Kiraz S, Krd N, Kayhan H, Yakut Y, Guler C. Validation of the Turkish version of the Oswestry Disability Index for patients with low back pain. Spine (Phila Pa 1976). 2004 Mar 1;29(5):581-5; discussion 585. doi: 10.1097/01.brs.0000113869.13209.03. PMID 15129077
- [Background] Wilby MJ, Best A, Wood E, Burnside G, Bedson E, Short H, Wheatley D, Hill-McManus D, Sharma M, Clark S, Baranidharan G, Price C, Mannion R, Hutchinson PJ, Hughes DA, Marson A, Williamson PR. Surgical microdiscectomy versus transforaminal epidural steroid injection in patients with sciatica secondary to herniated lumbar disc (NERVES): a phase 3, multicentre, open-label, randomised controlled trial and economic evaluation. Lancet Rheumatol. 2021 Mar 18;3(5):e347-e356. doi: 10.1016/S2665-9913(21)00036-9. eCollection 2021 May. PMID 33969319
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235
- [Background] Waddell G, Feder G, Lewis M. Systematic reviews of bed rest and advice to stay active for acute low back pain. Br J Gen Pract. 1997 Oct;47(423):647-52. PMID 9474831
- [Background] Verheijen EJA, Bonke CA, Amorij EMJ, Vleggeert-Lankamp CLA. Epidural steroid compared to placebo injection in sciatica: a systematic review and meta-analysis. Eur Spine J. 2021 Nov;30(11):3255-3264. doi: 10.1007/s00586-021-06854-9. Epub 2021 May 11. PMID 33974132
- [Background] Van Boxem K, Rijsdijk M, Hans G, de Jong J, Kallewaard JW, Vissers K, van Kleef M, Rathmell JP, Van Zundert J. Safe Use of Epidural Corticosteroid Injections: Recommendations of the WIP Benelux Work Group. Pain Pract. 2019 Jan;19(1):61-92. doi: 10.1111/papr.12709. Epub 2018 Jul 2. PMID 29756333
- [Background] Taspinar G, Angin E, Oksuz S. The effects of Pilates on pain, functionality, quality of life, flexibility and endurance in lumbar disc herniation. J Comp Eff Res. 2023 Jan;12(1):e220144. doi: 10.2217/cer-2022-0144. Epub 2022 Dec 1. PMID 36453667
- [Background] Soylu C, Kutuk B. Reliability and Validity of the Turkish Version of SF-12 Health Survey. Turk Psikiyatri Derg. 2022 Summer;33(2):108-117. doi: 10.5080/u25700. English, Turkish. PMID 35730511
- [Background] Skovrlj B, Gilligan J, Cutler HS, Qureshi SA. Minimally invasive procedures on the lumbar spine. World J Clin Cases. 2015 Jan 16;3(1):1-9. doi: 10.12998/wjcc.v3.i1.1. PMID 25610845
- [Background] Singh S, Kumar S, Chahal G, Verma R. Selective nerve root blocks vs. caudal epidural injection for single level prolapsed lumbar intervertebral disc - A prospective randomized study. J Clin Orthop Trauma. 2017 Apr-Jun;8(2):142-147. doi: 10.1016/j.jcot.2016.02.001. Epub 2016 Feb 22. PMID 28720990
- [Background] Sany SA, Mitsi M, Tanjim T, Rahman M. The effectiveness of different aerobic exercises to improve pain intensity and disability in chronic low back pain patients: a systematic review. F1000Res. 2023 Jul 18;11:136. doi: 10.12688/f1000research.75440.2. eCollection 2022. PMID 37854288
- [Background] Salik Sengul Y, Yilmaz A, Kirmizi M, Kahraman T, Kalemci O. Effects of stabilization exercises on disability, pain, and core stability in patients with non-specific low back pain: A randomized controlled trial. Work. 2021;70(1):99-107. doi: 10.3233/WOR-213557. PMID 34487008
- [Background] Rogers LJ, Bleetman D, Messenger DE, Joshi NA, Wood L, Rasburn NJ, Batchelor TJP. The impact of enhanced recovery after surgery (ERAS) protocol compliance on morbidity from resection for primary lung cancer. J Thorac Cardiovasc Surg. 2018 Apr;155(4):1843-1852. doi: 10.1016/j.jtcvs.2017.10.151. Epub 2017 Dec 19. PMID 29352586
- [Background] Rasouli MR, Rahimi-Movaghar V, Shokraneh F, Moradi-Lakeh M, Chou R. Minimally invasive discectomy versus microdiscectomy/open discectomy for symptomatic lumbar disc herniation. Cochrane Database Syst Rev. 2014 Sep 4;2014(9):CD010328. doi: 10.1002/14651858.CD010328.pub2. PMID 25184502
- [Background] Ozturk EC, Sacaklidir R, Sencan S, Gunduz OH. Caudal epidural steroid injection versus transforaminal ESI for unilateral S1 radiculopathy: a prospective, randomized trial. Pain Med. 2023 Aug 1;24(8):957-962. doi: 10.1093/pm/pnad041. PMID 37004169
- [Background] Ostelo RW, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, Bouter LM, de Vet HC. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 2008 Jan 1;33(1):90-4. doi: 10.1097/BRS.0b013e31815e3a10. PMID 18165753
- [Background] McCafferty B, Williams R. Epidural steroid injection technique. Tech Vasc Interv Radiol. 2024 Sep;27(3):100981. doi: 10.1016/j.tvir.2024.100981. Epub 2024 Aug 24. PMID 39490373
- [Background] Manchikanti L, Knezevic NN, Navani A, Christo PJ, Limerick G, Calodney AK, Grider J, Harned ME, Cintron L, Gharibo CG, Shah S, Nampiaparampil DE, Candido KD, Soin A, Kaye AD, Kosanovic R, Magee TR, Beall DP, Atluri S, Gupta M, Helm Ii S, Wargo BW, Diwan S, Aydin SM, Boswell MV, Haney BW, Albers SL, Latchaw R, Abd-Elsayed A, Conn A, Hansen H, Simopoulos TT, Swicegood JR, Bryce DA, Singh V, Abdi S, Bakshi S, Buenaventura RM, Cabaret JA, Jameson J, Jha S, Kaye AM, Pasupuleti R, Rajput K, Sanapati MR, Sehgal N, Trescot AM, Racz GB, Gupta S, Sharma ML, Grami V, Parr AT, Knezevic E, Datta S, Patel KG, Tracy DH, Cordner HJ, Snook LT, Benyamin RM, Hirsch JA. Epidural Interventions in the Management of Chronic Spinal Pain: American Society of Interventional Pain Physicians (ASIPP) Comprehensive Evidence-Based Guidelines. Pain Physician. 2021 Jan;24(S1):S27-S208. PMID 33492918
- [Background] Mallard F, Wong JJ, Lemeunier N, Cote P. Effectiveness of Multimodal Rehabilitation Interventions for Management of Cervical Radiculopathy in Adults: An Updated Systematic Review from the Ontario Protocol for Traffic Injury Management (Optima) Collaboration. J Rehabil Med. 2022 Aug 22;54:jrm00318. doi: 10.2340/jrm.v54.2799. PMID 35797062
- [Background] Luo X, George ML, Kakouras I, Edwards CL, Pietrobon R, Richardson W, Hey L. Reliability, validity, and responsiveness of the short form 12-item survey (SF-12) in patients with back pain. Spine (Phila Pa 1976). 2003 Aug 1;28(15):1739-45. doi: 10.1097/01.BRS.0000083169.58671.96. PMID 12897502
- [Background] Luan X, Tian X, Zhang H, Huang R, Li N, Chen P, Wang R. Exercise as a prescription for patients with various diseases. J Sport Health Sci. 2019 Sep;8(5):422-441. doi: 10.1016/j.jshs.2019.04.002. Epub 2019 Apr 18. PMID 31534817
- [Background] Kirwan JP, Sacks J, Nieuwoudt S. The essential role of exercise in the management of type 2 diabetes. Cleve Clin J Med. 2017 Jul;84(7 Suppl 1):S15-S21. doi: 10.3949/ccjm.84.s1.03. PMID 28708479
- [Background] Kim GE, Hong SJ, Kang SS, Ki HJ, Park JH. Epidural hematoma treated by aspiration after transforaminal epidural steroid injection - A case report. Anesth Pain Med (Seoul). 2021 Apr;16(2):184-190. doi: 10.17085/apm.20085. Epub 2021 Apr 9. PMID 33845549
- [Background] Kim DH, Yoon DM, Yoon KB. Incidence of intravascular injection and the spread of contrast media during S1 transforaminal epidural steroid injection by two approaches: anteroposterior vs oblique. Anaesthesia. 2015 Aug;70(8):975-84. doi: 10.1111/anae.13079. Epub 2015 Apr 7. PMID 25850817
- [Background] Kamanli A, Karaca-Acet G, Kaya A, Koc M, Yildirim H. Conventional physical therapy with lumbar traction; clinical evaluation and magnetic resonance imaging for lumbar disc herniation. Bratisl Lek Listy. 2010;111(10):541-4. PMID 21125798
- [Background] Jang JW, Lee DG, Park CK. Rationale and Advantages of Endoscopic Spine Surgery. Int J Spine Surg. 2021 Dec;15(suppl 3):S11-S20. doi: 10.14444/8160. PMID 34974417
- [Background] Hashemi M, Dadkhah P, Taheri M, Ghasemi M, Hosseinpour A, Farjam M. Patient-Reported Outcomes and Satisfaction after Cervical Epidural Steroid Injection for Cervical Radiculopathy. Galen Med J. 2019 Nov 3;8:e1478. doi: 10.31661/gmj.v8i0.1478. eCollection 2019. PMID 34466515
- [Background] Fornari M, Robertson SC, Pereira P, Zileli M, Anania CD, Ferreira A, Ferrari S, Gatti R, Costa F. Conservative Treatment and Percutaneous Pain Relief Techniques in Patients with Lumbar Spinal Stenosis: WFNS Spine Committee Recommendations. World Neurosurg X. 2020 Jun 23;7:100079. doi: 10.1016/j.wnsx.2020.100079. eCollection 2020 Jul. PMID 32613192
- [Background] Erol E, Yildiz A, Yildiz R, Apaydin U, Gokmen D, Elbasan B. Reliability and Validity of the Turkish Version of the Fremantle Back Awareness Questionnaire. Spine (Phila Pa 1976). 2019 May 1;44(9):E549-E554. doi: 10.1097/BRS.0000000000002909. PMID 30325886
- [Background] Costa F, Oertel J, Zileli M, Restelli F, Zygourakis CC, Sharif S. Role of surgery in primary lumbar disk herniation: WFNS spine committee recommendations. World Neurosurg X. 2024 Feb 23;22:100276. doi: 10.1016/j.wnsx.2024.100276. eCollection 2024 Apr. PMID 38496347
- [Background] Choi JY, Park SM, Kim HJ, Yeom JS. Recent Updates on Minimally Invasive Spine Surgery: Techniques, Technologies, and Indications. Asian Spine J. 2022 Dec;16(6):1013-1021. doi: 10.31616/asj.2022.0436. Epub 2022 Dec 27. PMID 36573300
- [Background] Cetingok H, Kanar M. Comparison of the eficacy of epidural steroid injection applied in cervical and lumbar regions. Agri. 2022 Jan;34(1):54-59. doi: 10.14744/agri.2022.46872. PMID 34988961
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Benyamin RM, Vallejo R, Wang V, Kumar N, Cedeno DL, Tamrazi A. Acute Epidural Hematoma Formation in Cervical Spine After Interlaminar Epidural Steroid Injection Despite Discontinuation of Clopidogrel. Reg Anesth Pain Med. 2016 May-Jun;41(3):398-401. doi: 10.1097/AAP.0000000000000397. PMID 27035463
- [Background] Badr M, Elkhawaga H, Fawaz K, Kasem M, Fayez E. Effects of Multimodal Physical Therapy on Pain, Disability, H-reflex, and Diffusion Tensor Imaging Parameters in Patients With Lumbosacral Radiculopathy Due to Lumbar Disc Herniation: A Preliminary Trial. Cureus. 2024 Jun 30;16(6):e63501. doi: 10.7759/cureus.63501. eCollection 2024 Jun. PMID 39081452
- [Background] Awadalla AM, Aljulayfi AS, Alrowaili AR, Souror H, Alowid F, Mahdi AMM, Hussain R, Alzahrani MM, Alsamarh AN, Alkhaldi EA, Alanazi RC. Management of Lumbar Disc Herniation: A Systematic Review. Cureus. 2023 Oct 29;15(10):e47908. doi: 10.7759/cureus.47908. eCollection 2023 Oct. PMID 38034203
- [Background] Alkhudari AM, Malk CS, Rahman A, Penmetcha T, Torres M. Epidural hematoma after routine epidural steroid injection. Surg Neurol Int. 2016 May 6;7:55. doi: 10.4103/2152-7806.181906. eCollection 2016. PMID 27213109
- [Background] Abubaker AK, Rabadi DK, Kassab M, Al-Qudah MA. Persistent Hiccups After Cervical Epidural Steroid Injection. Am J Case Rep. 2018 Apr 4;19:397-399. doi: 10.12659/ajcr.908536. PMID 29615600
- [Background] Abenhaim L, Rossignol M, Valat JP, Nordin M, Avouac B, Blotman F, Charlot J, Dreiser RL, Legrand E, Rozenberg S, Vautravers P. The role of activity in the therapeutic management of back pain. Report of the International Paris Task Force on Back Pain. Spine (Phila Pa 1976). 2000 Feb 15;25(4 Suppl):1S-33S. doi: 10.1097/00007632-200002151-00001. No abstract available. PMID 10707404